CLINICAL TRIAL: NCT02436863
Title: Influence of Laminoplasty and Internal Fixation on Vertebral Stability After Cervical, Thoracic and Lumbar Laminectomy for Tumor Resection
Brief Title: Influence of Laminoplasty and Internal Fixation on Vertebral Stability After Laminectomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Southern Medical University, China (Other)
Responsible Party: Principal Investigator, Yuntao Lu, Professor, Southern Medical University, China
Other Study IDs: SMU-spine-1
Record Dates: First submitted 2015-05-04; First posted 2015-05-07 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Disorders Following Clinical Procedure
Keywords: Laminectomy; Laminoplasty; Internal fixation; deformity
MeSH Terms: conditions — Congenital Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Surgical perfomance (Laminoplasty): After the lesions inside the spinal canal were surgical removed by laminectomy, the lamina and spinous process were replanted with titanium plates and screws.
  Interventions: Procedure: Surgical performance
- Surgical perfomance (Internal fixation): After the lesions inside the spinal canal were surgical removed by laminectomy, the pedicle screws (Thoracic and lumbar vertebra) or lateral mass (Cervical vertebra) and sticks were used for internal fixation.
  Interventions: Procedure: Surgical performance

INTERVENTIONS:
Procedure: Surgical performance — Two different surgical performances

SUMMARY:
The lesion located inside the spinal canal caused big trouble for clinical treatment. Traditional laminectomy will destroy the biomechanics and influent the vertebral stability, which might cause kyphosis or other deformity. So in some centers, neurosurgeries praised laminoplasty to make the intactness of posterior column. They thought the laminoplasty can maintain the vertebral stability, and meanwhile the range of motion won't change so much. However, some other scholars thought laminoplasty had no helps for stability because of the pseudarthrosis. They preferred screw and stick system for internal fixation. And we did meet several patients after laminectomy suffered with spinal deformity. So we thought it is necessary for investigating the benefit of patients from laminoplasty and internal fixation.

DETAILED DESCRIPTION:
After laminectomy for removal of the cervical, thoracic and lumbar lesions, the recruited cases were randomly divided into two groups.

1. The cases in group of laminoplasty, the lamina and spinous process was replanted to maintain the anatomical intactness of spinal canal.
2. On the other hand, the cases in internal fixation group, the pedicle screws were implanted, and tickets were used to complete the internal fixation.

During 3 years follow up, the vertebral deformity and the range of motion were investigated and evaluated. And in the meantime, the patient's age will also be analyzed to detect it's influence for the prognosis.

ELIGIBILITY:
Inclusion Criteria:

- 1. Adult patients (>=18 years) were enrolled. 2. The patients suffered with lesion inside the spinal canal, who underwent laminectomy to remove the lesion.

3. Pathology proved benign lesion. 4. Health condition of patients (KPS) >= 70.

Exclusion Criteria:

* 1. Children cases (<18 years) were excluded.
* 2.The cases with pathological malignant tumors were excluded from this study.
* 3. KPS of patients < 70.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Adult patients (>18 years) were enrolled.
  2. The patients suffered with lesion inside the spinal canal, who underwent laminectomy to remove the lesion.
  3. The cases with pathological malignant tumors were excluded from this study.
  4. Health condition of patients (KPS) > 70.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2015-01; Primary Completion 2018-12 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Vertebral deformity | 3 years

SECONDARY OUTCOMES:
The influence of age on the vertebral deformity | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Yuntao Lu, M.D., Ph.D, Principal Investigator — Nanfang neurosurgery research institution
Locations (1):
- Nan fang hospital, Southern medical university, Guangzhou, Guangdong, China